CLINICAL TRIAL: NCT01075178
Title: Palivizumab (Synagis®) Post-marketing Surveillance Cohort Study in Children < 24 Months of Age With Hemodynamically Significant Congenital Heart Disease
Brief Title: Retrospective Palivizumab Study in Children With Hemodynamically Significant Congenital Heart Disease
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Responsible Party: Andrew L. Campbell, M.D., Medical Director, Abbott
Other Study IDs: M03-681
Record Dates: First submitted 2010-02-23; First posted 2010-02-25 (Estimated); Results first posted 2011-02-24 (Estimated); Last update posted 2011-03-23 (Estimated); Status verified 2011-03

CONDITIONS: Severe Respiratory Syncytial Virus Infection
Keywords: Infection; Arrhythmia; Death; Palivizumab; Safety; Hemodynamically Significant Congenital Heart Disease; Pediatric; Observational
MeSH Terms: conditions — Respiratory Syncytial Virus Infections; Infections; Arrhythmias, Cardiac; Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Palivizumab-treated subjects (CASES): HSCHD infants, <2 yrs old at first dose of palivizumab
- Non-palivizumab-treated subjects (CONTROLS): HSCHD infants, <2 yrs old that did not receive palivizumab

SUMMARY:
Retrospective medical record review study of specific adverse events in children with congenital heart disease who received palivizumab for prophylaxis of serious respiratory syncytial virus infection and control subjects that did not receive palivizumab

DETAILED DESCRIPTION:
This is an observational, non-interventional, retrospective cohort study of infants with hemodynamically significant congenital heart disease (HSCHD) who were less than 24 months of age when the first dose of palivizumab was administered (CASES), and infants who were diagnosed with hemodynamically significant congenital heart disease but did not receive palivizumab in a historical respiratory syncytial virus (RSV) season during the first 24 months of life (CONTROLS). CASES are matched to CONTROLS based on RSV season, age, type of cardiac lesion, and type of prior corrective cardiac surgery. Subject medical records are reviewed for occurrences of the clinical end points of infection, arrhythmia, and/or death that meet criteria for serious adverse events. The groups will be compared for number and percent of subjects who experience these primary serious adverse events (both individually and collectively) during a defined 8-month chart review period.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have documented hemodynamically significant congenital heart disease (Note: Children with uncomplicated small atrial or ventricular septal defects or patent ductus arteriosus are not eligible).
2. Subject must have unoperated or partially corrected congenital heart disease.
3. Subject must have received at least one dose of palivizumab for prophylaxis during the Respiratory Syncytial Virus season - September 1 through April 30 (CASES), or would have been considered eligible for palivizumab prophylaxis (CONTROLS).
4. Subject must be < 24 months of age at the time of the first dose of palivizumab prophylaxis (CASES) or < 32 months of age at the end of the assigned Respiratory Syncytial Virus season in which they would have been eligible to receive palivizumab if the drug had been approved in the European Union (CONTROLS).
5. Subject's parent, guardian, or legal representative has voluntarily signed and dated a Release of Information Form to allow the review of medical records and collection of pertinent study data.

Exclusion Criteria:

1. Subject was contraindicated for treatment with palivizumab according to the current European product label.
2. Subject had full correction of Congenital Heart Disease.
3. Subject received palivizumab before approval for use in Congenital Heart Disease (CASES), or subject received palivizumab at any time (CONTROLS).
4. Subject has already been included in this study in a prior Respiratory Syncytial Virus season.

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children less than 24 months of age with hemodynamically significant congenital heart disease
Sampling Method: Non-Probability Sample
Enrollment: 2036 (Actual)
Dates: Start 2006-07; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Campbell, MD, Study Director — Medical Director, Abbott Laboratories
Locations (37):
- Austria (3):
  - Site Reference ID/Investigator# 6263, Linz
  - Site Reference ID/Investigator# 7956, Vienna
  - Site Reference ID/Investigator# 9403, Vienna
- Belgium (3):
  - Site Reference ID/Investigator# 17821, Brussels
  - Site Reference ID/Investigator# 18602, Ghent
  - Site Reference ID/Investigator# 18601, Leuven
- France (4):
  - Site Reference ID/Investigator# 6244, Nantes
  - Site Reference ID/Investigator# 6261, Paris
  - Site Reference ID/Investigator# 6245, Paris
  - Site Reference ID/Investigator#6260, Reims
- Germany (9):
  - Site Reference ID/Investigator# 6280, Bad Oeynhausen
  - Site Reference ID/Investigator# 9621, Berlin
  - Site Reference ID/Investigator# 16361, Braunschweig
  - Site Reference ID/Investigator# 6283, Duisburg
  - Site Reference ID/Investigator# 6272, Essen
  - Site Reference ID/Investigator# 6271, Göttingen
  - Site Reference ID/Investigator# 8277, Munich
  - Site Reference ID/Investigator# 11182, Rostock
  - Site Reference ID/Investigator# 6249, Sankt Augustin
- Italy (5):
  - Site Reference ID/Investigator# 6274, Campobasso
  - Site Reference ID/Investigator# 6276, Florence
  - Site Reference ID/Investigator# 4703, Naples
  - Site Reference ID/Investigator# 4910, Padua
  - Site Reference ID/Investigator# 14681, Roma
- Site Reference ID/Investigator# 14802, Trondheim, Norway
- Poland (4):
  - Site Reference ID/Investigator# 6275, Bydgoszcz
  - Site Reference ID/Investigator# 13102, Katowice
  - Site Reference ID/Investigator# 6270, Krakow
  - Site Reference ID/Investigator# 12222, Warsaw
- Site Reference ID/Investigator# 14682, Ljubljana, Slovenia
- Spain (4):
  - Site Reference ID/Investigator# 5372, A Coruña
  - Site Reference ID/Investigator# 15381, Madrid
  - Site Reference ID/Investigator# 15702, Madrid
  - Site Reference ID/Investigator# 15261, Santiago de Compostela
- United Kingdom (3):
  - Site Reference ID/Investigator# 6282, Belfast
  - Site Reference ID/Investigator# 13941, Bristol
  - Site Reference ID/Investigator# 5023, London

REFERENCES:
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/drugInfo.cfm?id=23151&CFID

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Infants diagnosed with hemodynamically significant congenital heart disease who were less than 24 months of age when first dosed with palivizumab (CASES) were compared for the occurrence of serious adverse events over an 8-month chart review period with matched infants who did not receive palivizumab during the first 24 months of life (CONTROLS).
Period: Subject Matching
Arm/Group | Palivizumab-treated Subjects (CASES) | Non-palivizumab-treated Subjects (CONTROLS)
Started | 1148 (eligible for matching) | 1421 (eligible for matching)
Completed | 1018 (subjects matched) | 1018 (subjects matched)
Not Completed | 130 | 403
Not completed — eligible but not matched | 130 | 403
Period: Subject Chart Review
Arm/Group | Palivizumab-treated Subjects (CASES) | Non-palivizumab-treated Subjects (CONTROLS)
Started | 1018 (subjects matched) | 1018 (subjects matched)
Completed | 1009 (subjects in full analysis set) | 1009 (subjects in full analysis set)
Not Completed | 9 | 9
Not completed — died before chart review period | 0 | 2
Not completed — no data collected due to site closure | 3 | 4
Not completed — matched partner excluded (reasons above) | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Palivizumab-treated Subjects (CASES) | Non-palivizumab-treated Subjects (CONTROLS) | Total
Number analyzed (Participants) | 1009 | 1009 | 2018
Age Categorical [Number; unit: participants]
  <=6 months | 651 | 656 | 1307
  >6 months | 358 | 353 | 711
Age Continuous [Mean (Standard Deviation); unit: months] | 5.4 (4.91) | 5.4 (5.05) | 5.4 (4.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 437 | 462 | 899
  Male | 572 | 547 | 1119
Region of Enrollment [Number; unit: participants]
  France | 188 | 211 | 399
  Slovenia | 16 | 20 | 36
  Spain | 284 | 170 | 454
  Poland | 36 | 242 | 278
  Belgium | 77 | 115 | 192
  Austria | 96 | 53 | 149
  Norway | 12 | 7 | 19
  Germany | 97 | 90 | 187
  United Kingdom | 92 | 59 | 151
  Italy | 111 | 42 | 153
Cardiac lesion [Number; unit: participants]
  Cyanotic | 488 | 487 | 975
  Acyanotic | 521 | 522 | 1043
Corrective cardiac surgery [Number; unit: participants]
  None | 484 | 485 | 969
  Partially corrected congenital heart disease | 525 | 521 | 1046
  Fully corrected congenital heart disease | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Comparison Between CASES and CONTROLS of the Occurrence of Specific Clinical Outcomes of Serious Infection, Serious Arrhythmia and/or Death
Description: The number of subjects who experienced at least 1 event of infection, arrhythmia, or death meeting any of the criteria for a serious adverse event
Time Frame: 8-month chart review period in CASES and CONTROLS
Population: The population analyzed included the full analysis set.
Measure: Number; unit: participants
Arm/Group | Palivizumab-treated Subjects (CASES) | Non-palivizumab-treated Subjects (CONTROLS)
Number analyzed (Participants) | 1009 | 1009
participants | 303 | 349
Statistical Analysis 1: Comparison: Palivizumab-treated Subjects (CASES) vs Non-palivizumab-treated Subjects (CONTROLS); The null hypothesis was that the odds ratio was greater than or equal to 2. The planned sample size of 2000 participants (1000 participants in each group) provided greater than 90% power to determine non-inferiority based on the odds ratio less than 2; Test type: Non-Inferiority or Equivalence — Non-inferiority was assessed with a 95% 1-sided confidence interval for which the upper bound of the difference in the event rates (CASES minus CONTROLS) will correspond to an odds ratio less than 2 (that is, the odds ratio calculated at the upper confidence bound of the difference in event rates will be less than 2); exact binomial; Observed odds ratio = 0.81, 95% CI 1-sided [upper limit 0.96] — Result provided for "95% Confidence Interval (1-Sided)" is the odds ratio calculated at the upper bound of the 1-sided 95% confidence interval for the difference in event rates (CASES minus CONTROLS)

2. Primary Outcome: Comparison Between CASES and CONTROLS of the Occurrence of Specific Clinical Outcomes of Serious Infection.
Description: The number of subjects who experienced at least 1 event of infection meeting any of the criteria for a serious adverse event
Time Frame: 8-month chart review period in CASES and CONTROLS
Population: The population analyzed included the full analysis set.
Measure: Number; unit: participants
Arm/Group | Palivizumab-treated Subjects (CASES) | Non-palivizumab-treated Subjects (CONTROLS)
Number analyzed (Participants) | 1009 | 1009
participants | 281 | 329
Statistical Analysis 1: Comparison: Palivizumab-treated Subjects (CASES) vs Non-palivizumab-treated Subjects (CONTROLS); [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; exact binomial; Observed odds ratio = 0.80, 95% CI 1-sided [upper limit 0.95] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Comparison Between CASES and CONTROLS of the Occurrence of Specific Clinical Outcomes of Serious Arrhythmia
Description: The number of subjects who experienced at least 1 event of arrhythmia meeting any of the criteria for a serious adverse event
Time Frame: 8-month chart review period in CASES and CONTROLS
Population: The population analyzed included the full analysis set.
Measure: Number; unit: participants
Arm/Group | Palivizumab-treated Subjects (CASES) | Non-palivizumab-treated Subjects (CONTROLS)
Number analyzed (Participants) | 1009 | 1009
participants | 41 | 39
Statistical Analysis 1: Comparison: Palivizumab-treated Subjects (CASES) vs Non-palivizumab-treated Subjects (CONTROLS); [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; exact binomial; Observed odds ratio = 1.05, 95% CI 1-sided [upper limit 1.64] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Comparison Between CASES and CONTROLS of the Occurrence of Specific Clinical Outcomes of Death
Description: The number of subjects who died
Time Frame: 8-month chart review period in CASES and CONTROLS
Population: The population analyzed included the full analysis set.
Measure: Number; unit: participants
Arm/Group | Palivizumab-treated Subjects (CASES) | Non-palivizumab-treated Subjects (CONTROLS)
Number analyzed (Participants) | 1009 | 1009
participants | 9 | 10
Statistical Analysis 1: Comparison: Palivizumab-treated Subjects (CASES) vs Non-palivizumab-treated Subjects (CONTROLS); [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; exact binomial; Observed odds ratio = 0.90, 95% CI 1-sided [upper limit 2.19] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: 8-month chart review period
Description: Only serious adverse events of infection, arrhythmia, and death were collected and assessed as part of the study; other (non-serious) adverse events were not collected or assessed.
Arm/Group | Palivizumab-treated Subjects (CASES) | Non-palivizumab-treated Subjects (CONTROLS)
Serious Adverse Events (participants affected / at risk) | 303/1009 | 349/1009
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Palivizumab-treated Subjects (CASES) (N=1009) | Non-palivizumab-treated Subjects (CONTROLS) (N=1009)
Arrhythmia (Cardiac disorders) | 4 | 8
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 0
Atrial tachycardia (Cardiac disorders) | 1 | 2
Atrioventricular block (Cardiac disorders) | 4 | 3
Atrioventricular block complete (Cardiac disorders) | 1 | 4
Atrioventricular block second degree (Cardiac disorders) | 3 | 0
Bradycardia (Cardiac disorders) | 2 | 5
Cardiac arrest (Cardiac disorders) | 1 | 2
Cardiac failure (Cardiac disorders) | 1 | 5
Extrasystoles (Cardiac disorders) | 0 | 1
Myocarditis (Cardiac disorders) | 0 | 1
Nodal arrhythmia (Cardiac disorders) | 6 | 7
Nodal rhythm (Cardiac disorders) | 4 | 0
Pericarditis (Cardiac disorders) | 1 | 1
Sinus arrhythmia (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 10 | 5
Tachycardia (Cardiac disorders) | 1 | 2
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Congenital infection (Congenital, familial and genetic disorders) | 1 | 0
Congenital pneumonia (Congenital, familial and genetic disorders) | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Enterocolitis (Gastrointestinal disorders) | 0 | 4
Gastritis (Gastrointestinal disorders) | 1 | 0
Necrotising colitis (Gastrointestinal disorders) | 0 | 1
Peritonitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 1
Hepatitis toxic (Hepatobiliary disorders) | 0 | 1
Acarodermatitis (Infections and infestations) | 1 | 0
Acinetobacter infection (Infections and infestations) | 0 | 1
Adenovirus infection (Infections and infestations) | 1 | 1
Anal abscess (Infections and infestations) | 0 | 1
Bacillus infection (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 5 | 0
Bacterial infection (Infections and infestations) | 3 | 3
Bronchiolitis (Infections and infestations) | 47 | 40
Bronchitis (Infections and infestations) | 19 | 38
Bronchitis viral (Infections and infestations) | 0 | 1
Bronchopneumonia (Infections and infestations) | 1 | 22
Candida sepsis (Infections and infestations) | 0 | 1
Candidiasis (Infections and infestations) | 0 | 1
Candiduria (Infections and infestations) | 0 | 1
Catheter sepsis (Infections and infestations) | 0 | 1
Central line infection (Infections and infestations) | 2 | 1
Clostridial infection (Infections and infestations) | 0 | 1
Croup infectious (Infections and infestations) | 2 | 1
Dermatitis infected (Infections and infestations) | 0 | 1
Ear infection (Infections and infestations) | 3 | 2
Endocarditis (Infections and infestations) | 1 | 0
Endicarditis enterococcal (Infections and infestations) | 0 | 1
Enterobacter sepsis (Infections and infestations) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 1 | 0
Exanthema subitum (Infections and infestations) | 0 | 3
Eye infection (Infections and infestations) | 0 | 1
Fungal infection (Infections and infestations) | 1 | 0
Gastric infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 42 | 36
Gastroenteritis adenovirus (Infections and infestations) | 1 | 0
Gastroenteritis norovirus (Infections and infestations) | 8 | 0
Gastroenteritis rotavirus (Infections and infestations) | 3 | 9
Gastroenteritis salmonella (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 1
Gastrointestinal infection (Infections and infestations) | 2 | 2
Haemophilus infection (Infections and infestations) | 1 | 1
Incision site abscess (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 8 | 15
Influenza (Infections and infestations) | 1 | 0
Klebsiella infection (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 3 | 3
Lobar pneumonia (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 7 | 6
Lower respiratory tract infection viral (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 9 | 7
Mediastinitis (Infections and infestations) | 2 | 1
Meningitis (Infections and infestations) | 1 | 0
Metapneumovirus infection (Infections and infestations) | 1 | 0
Moraxella infection (Infections and infestations) | 1 | 1
Nasopharyngitis (Infections and infestations) | 0 | 2
Nosocomial infection (Infections and infestations) | 5 | 1
Oral candidiasis (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0
Orchitis (Infections and infestations) | 0 | 1
Otitis externa (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 3 | 9
Otitis media acute (Infections and infestations) | 1 | 1
Parainfluenza virus infection (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 2 | 5
Pneumococcal sepsis (Infections and infestations) | 0 | 1
Pneumocystitis jiroveci infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 30 | 38
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pneumonia klebsiella (Infections and infestations) | 1 | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 2
Pneumonia streptococcal (Infections and infestations) | 1 | 1
Pneumonia viral (Infections and infestations) | 1 | 0
Post procedural infection (Infections and infestations) | 3 | 14
Post procedural pneumonia (Infections and infestations) | 1 | 0
Post procedural sepsis (Infections and infestations) | 0 | 2
Postoperative wound infection (Infections and infestations) | 6 | 4
Pseudomonas infection (Infections and infestations) | 3 | 3
Pyelonephritis (Infections and infestations) | 2 | 1
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 5 | 17
Respiratory syncytial virus infection (Infections and infestations) | 4 | 5
Respiratory tract infection (Infections and infestations) | 19 | 19
Respiratory tract infection bacterial (Infections and infestations) | 1 | 1
Respiratory tract infection viral (Infections and infestations) | 3 | 2
Rhinitis (Infections and infestations) | 2 | 2
Rotavirus infection (Infections and infestations) | 1 | 4
Sepsis (Infections and infestations) | 23 | 24
Septic shock (Infections and infestations) | 0 | 2
Serratia infection (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 2 | 3
Staphylococcal sepsis (Infections and infestations) | 2 | 2
Stenotrophomonas infection (Infections and infestations) | 1 | 0
Systemic candida (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 2 | 2
Tracheitis (Infections and infestations) | 2 | 5
Tracheobronchitis (Infections and infestations) | 1 | 0
Tracheostomy infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 25 | 23
Urinary tract infection (Infections and infestations) | 31 | 36
Urinary tract infection bacterial (Infections and infestations) | 2 | 0
Urosepsis (Infections and infestations) | 1 | 0
Varicella (Infections and infestations) | 2 | 1
Viral infection (Infections and infestations) | 8 | 3
Viral tonsillitis (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 5 | 3
Wound infection fungal (Infections and infestations) | 1 | 0
Wound infection staphylococcal (Infections and infestations) | 0 | 1
Cardiac pacemaker malfunction (Injury, poisoning and procedural complications) | 1 | 0
Clostridium difficile toxin test (Investigations) | 1 | 0
Respiratory syncytial virus test positive (Investigations) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Febrile convulsion (Nervous system disorders) | 2 | 0
Syncope (Nervous system disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hangnail (Skin and subcutaneous tissue disorders) | 0 | 1
Cardiogenic shock (Cardiac disorders) | 1 | 0
Congestive cardiomyopathy (Cardiac disorders) | 1 | 0
Heart disease congenital (Congenital, familial and genetic disorders) | 1 | 0
Hypoplastic left heart syndrome (Congenital, familial and genetic disorders) | 1 | 0
Heart transplant rejection (Immune system disorders) | 1 | 0
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemodynamic instability (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Only serious adverse events of infection and arrhythmia as well as deaths were collected in this study. The criterion for non-inferiority was not met for death, most likely because the reported mortality rates were lower than expected in both groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.